CLINICAL TRIAL: NCT00321217
Title: Pharmacogenomics of Anti-TNF Treatment in Patients With Rheumatoid Arthritis
Brief Title: Pharmacogenomics of Anti-TNF (Anti-tumor Necrosis Factor) Treatment in Patients With Rheumatoid Arthritis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: pharmacogenomics of anti-TNF
Record Dates: First submitted 2006-05-02; First posted 2006-05-03 (Estimated); Last update posted 2012-08-16 (Estimated); Status verified 2011-11

CONDITIONS: Rheumatoid Arthritis
Keywords: rheumatoid arthritis; pharmacogenetics; anti-TNF; high throughput genotyping
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The main aim of this study is to identify genetic markers (at DNA and RNA level) which are involved in the response to treatment with monoclonal antibodies against TNF in patients with rheumatoid arthritis.

DETAILED DESCRIPTION:
Rheumatoid Arthritis (RA) is a severe inflammatory disease and genetic factors are known to play an important role in its pathogenesis. Genetic factors are also involved in determining the prognosis of RA. Identifying the genetic factors that predispose to mild or aggressive RA is not easy and up to now only a few of these factors -like certain HLA-DR species- are known.

The Rheumatology department of the Radboud University Nijmegen Medical Centre (RUNMC) has collected a unique inception cohort of over 500 patients with RA, that have been followed from an early stage of disease for up to 10 years with detailed measurements of disease activity, joint damage and other characteristics of disease progression.

In this project we use this patient group to study polymorphisms in a large battery of genes for their effect on RA disease activity/progression.

ELIGIBILITY:
Inclusion Criteria:

* Patients with RA according to the ACR criteria who are treated with monoclonal anti-TNF antibodies.

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with RA according to the ACR criteria who are treated with monoclonal anti-TNF antibodies.
Sampling Method: Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2004-05; Primary Completion 2013-11 (Estimated); Study Completion 2014-04 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: M. J. Coenen, PhD, Principal Investigator — Radboud University Medical Center
Locations (3):
- Netherlands (3):
  - Rijnstate, Arnhem
  - Radboud University Nijmegen Medical Centre, Nijmegen
  - St Maartenskliniek, Nijmegen